CLINICAL TRIAL: NCT07254260
Title: Photodynamic Therapy (PDT) and Postendodontic Pain
Brief Title: Photodynamic Therapy and Post-Endodontic Pain in Undergraduate-Performed Treatments
Acronym: PDT
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Ayfer Atav, Assoc Prof, Atlas University
Other Study IDs: E-22686390-050.99-78516; E-22686390-050.99-78516 (Other: Istanbul Atlas University Non-Interventional Scientific Research Ethics Committee)
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pulpitis
Keywords: Postendodontic pain
MeSH Terms: conditions — Pulpitis | interventions — Photochemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conventional Final Irrigation Without Activation (Control Group): The final irrigation protocol consisted of sequential rinses with saline, 17% ethylenediaminetetraacetic acid (EDTA; Wizard, Turkey), and distilled water and 2.5% sodium hypochlorite (NaOCl; Wizard, Turkey), which was activated during this step, followed by a final flush with saline solution.
  Interventions: Device: Photodynamic Therapy
- Brief Title: The Effect of Photodynamic Therapy on Post-Endodontic Pain in Treatments P: Following completion of standard chemomechanical preparation and photodynamic therapy (PDT) was performed using the Easyinsmile Photodynamic PDT 630 System (Easyinsmile Co., Ltd., Changsha, Hunan, China). A low-range photosensitizer solution (Easyinsmile Photosensitizer, methylene blue-based formulation, λ_max = 630 nm) was delivered into each prepared root canal using the dedicated delivery syringe tip provided with the photosensitizer, ensuring precise, controlled placement of the agent while minimizing the risk of apical extrusion. The Easyinsmile endo-type light guard tip (diameter: 200 µm; emission wavelength: 630 ± 10 nm; optical power density: approximately 100 mW/cm²) was inserted into the canal. Photoactivation was then performed for 30 seconds per canal (10-second periods x 3).
  Interventions: Device: Photodynamic Therapy

INTERVENTIONS:
Device: Photodynamic Therapy — the Easyinsmile endo-type light guard tip (diameter: 200 µm; emission wavelength: 630 ± 10 nm; optical power density: approximately 100 mW/cm²) was inserted into the canal. Photoactivation was then performed for 30 seconds per canal (10 second periods x 3).

SUMMARY:
To compare the intensity and trajectory of postoperative pain (0-72 hours) between (A) a conventional final irrigation protocol without activation and (B) a PDT-augmented final disinfection in mandibular molars and premolars.

DETAILED DESCRIPTION:
This retrospective controlled clinical cohort study investigated the effects of photodynamic therapy (PDT) on post-endodontic pain in mandibular molars and premolars treated by undergraduate students. Eligible patients were selected from the Istanbul Atlas University Faculty of Dentistry clinics. Inclusion criteria encompassed adult patients requiring endodontic treatment in posterior teeth, without systemic contraindications or signs of acute apical abscess.

Participants were assigned to one of two groups:

(A) conventional final irrigation without activation (control), and (B) PDT-augmented final disinfection (experimental).

All treatments were performed by undergraduate dental students under faculty supervision. Root canals were shaped using a standardized rotary instrumentation protocol. In both groups, final irrigation included 2.5% sodium hypochlorite (NaOCl), followed by 17% EDTA for smear layer removal.

In the experimental group, after completion of the same irrigation regimen, a methylene blue photosensitizer was introduced into the canal and allowed to remain for 60 seconds. The dye was subsequently activated using an intra-canal diode laser fiber for 60 seconds per canal, following manufacturer instructions for photodynamic therapy. All canals were obturated at the second visit using the single-cone technique.

Postoperative pain was measured using a visual analog scale (VAS) at 6, 24, 48, and 72 hours after treatment. Additional variables such as analgesic consumption, incidence of flare-ups, unscheduled visits, and the time required to achieve a pain-free state were also recorded. This study aimed to determine whether adjunctive PDT could reduce early post-endodontic pain in treatments performed by undergraduate practitioners.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-60 years Patients requiring primary endodontic treatment of posterior teeth (premolars or molars) Patients without systemic diseases Patients treated at the Istanbul Atlas University Faculty of Dentistry student clinic Teeth with no intraoperative complications (no perforation, no instrument separation, no ledge formation) Treatments completed with either photodynamic therapy (PDT) activation or no activation (control group)

Exclusion Criteria:

Teeth with previous root canal treatment Teeth with open apices Presence of severe periodontal disease Incomplete clinical or radiographic records Patients with systemic conditions that may influence postoperative pain perception Any intraoperative complications during treatment (perforation, ledge, instrument separation, etc.) Presence of acute apical abscess

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged 18-60 years who received primary endodontic treatment of mandibular premolars or molars at the Istanbul Atlas University Faculty of Dentistry student clinic. All treatments were performed by undergraduate dental students under supervision. Eligible patients had no systemic diseases and presented with teeth requiring primary root canal therapy without intraoperative complications.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity (Visual Analog Scale - VAS) | Time Frame: 6, 24, 48, and 72 hours after treatment Unit of Measure: VAS score (0-10)
  Postoperative pain will be assessed using a 10-cm Visual Analog Scale (VAS), where 0 represents "no pain" and 10 represents "worst pain imaginable." Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Analgesic Consumption (Number of Tablets Taken) | Up to 72 hours after treatment
  The number of analgesic tablets consumed by each participant during the postoperative period will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayfer ATAV ATEŞ, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chiniforush N, Pourhajibagher M, Shahabi S, Kosarieh E, Bahador A. Can Antimicrobial Photodynamic Therapy (aPDT) Enhance the Endodontic Treatment? J Lasers Med Sci. 2016 Spring;7(2):76-85. doi: 10.15171/jlms.2016.14. Epub 2016 Mar 27. PMID 27330702